CLINICAL TRIAL: NCT00577408
Title: Behavioral Naltrexone Therapy (BNT) for Promoting Adherence to Oral Naltrexone (BNT-oral) vs Extended Release Injectable Depot Naltrexone (Depot-BNT); a Randomized Trial
Brief Title: Behavioral Naltrexone Therapy for Promoting Adherence to Oral Naltrexone vs Extended Release Injectable Depot Naltrexone
Acronym: Depot-BNT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #5307; R01DA010746 (NIH)
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Opiate Dependence; Heroin Dependence
Keywords: Opiate Dependence; Heroin Dependence; Naltrexone
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Depot Naltrexone (Experimental): Depot Naltrexone. Vivitrol (380 mg)given monthly
  Interventions: Drug: depot naltrexone
- Oral Naltrexone (Active Comparator): Oral Naltrexone. For patients assigned to BNT-Oral, administration is clinic-based for at least the first two weeks, and doses are 50mg, 100mg, or 150mg, depending on whether one, two or three days will elapse before the next visit (typically 100 mg on Monday and Wednesday and 150 mg on Friday).
  Interventions: Drug: Oral Naltrexone

INTERVENTIONS:
Drug: depot naltrexone — On the afternoon of Day 7, patients assigned to Depot-BNT receive an intramuscular injection of Vivitrol (380 mg) in one buttock. The patient spends the night of Day 7 in the hospital and is discharged on the morning of Day 8. Each injection contains 192 mg of naltrexone. The double dose (384 mg) is what was found to produce optimal blockade and outcome in preliminary work. During the subsequent 6-month course of outpatient treatment, patients are dosed with two injections (384 mg total) of depot naltrexone at monthly intervals (weeks 4, 8, 12, 16, 20).
  Other Names: Vivitrol
  Arms: Depot Naltrexone
Drug: Oral Naltrexone — For patients assigned to BNT-Oral, administration is clinic-based for at least the first two weeks, and doses are 50mg, 100mg, or 150mg, depending on whether one, two or three days will elapse before the next visit (typically 100 mg on Monday and Wednesday and 150 mg on Friday). The ultimate goal with BNT-Oral is for patients to take naltrexone (50 mg per day) on their own at home under supervision of their significant other/monitor.
  Other Names: Revia
  Arms: Oral Naltrexone

SUMMARY:
In pilot study now proposed, we plan to randomly assign 60 opioid dependent patients to the new model, Depot-BNT, or to BNT plus oral naltrexone for a 6-month trial. This will provide initial clinical experience with the new Depot-BNT treatment model, while providing a rigorous test of whether Depot-BNT produces superior treatment outcome, compared to our best behavioral platform for oral naltrexone (BNT).

The following aims will be addressed:

Specific Aim #1: To test whether Depot-BNT increases retention in treatment and improves drug use outcome (urine-confirmed abstinent weeks) compared to our established model of BNT with oral naltrexone (BNT-Oral), and to explore whether Depot-BNT (vs BNT-Oral) improves key secondary outcomes including dysphoria, HIV risk behavior, and social functioning.

Specific Aim #2: To explore predictors of outcome on Depot-BNT, and mechanisms of attrition, in order to optimize Depot-BNT prior to further testing.

DETAILED DESCRIPTION:
The clinical trial now proposed will provide an initial test of the feasibility and efficacy of the newly adapted version of Behavioral Naltrexone Therapy for Depot Naltrexone (Depot-BNT). Treatment-seeking opiate-dependent patients will be admitted for inpatient detoxification and induction onto oral naltrexone. Those who are successfully inducted will be randomly assigned for a six month trial to one of two conditions: 1) Behavioral Naltrexone Therapy for Depot Naltrexone (Depot-BNT) (N = 30), with the first dose of depot naltrexone administered prior to discharge from hospital with monthly doses thereafter; or 2) Behavioral Naltrexone Therapy as previously developed for promoting compliance with daily oral naltrexone (BNT-Oral) (N = 30). All patients in both groups will be asked to attend twice weekly outpatient therapy sessions over a six month course. This design will provide a test of whether Depot-BNT produces superior treatment retention and drug use outcome in comparison to our established behavioral platform for oral naltrexone, while providing experience upon which to base revisions of Depot-BNT prior to embarking upon further Stage 2 testing. Treatment will take place at the same sites as for our prior studies: (1) the General Clinical Research Unit (GCRU) of New York State Psychiatric Institute (NYSPI) and (2) the Substance Treatment and Research Service (STARS) of the Division on Substance Abuse at NYSPI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60.
2. Meets DSM-IV criteria for current opiate dependence disorder of at least six months duration, supported by a positive urine for opiates and a positive naloxone challenge test if the diagnosis is unclear. If participating as an outpatient only, recent opiate dependence must be confirmed by clinical history and/or communication with former treatment provider.
3. Seeking treatment for heroin dependence.
4. Able to give informed consent.

Exclusion Criteria:

1. Methadone maintenance treatment or regular use of illicit methadone (> 30 mg per week).
2. Maintenance on, or regular use of buprenorphine or other long-acting narcotic agonists.
3. Pregnancy, lactation, or failure in a sexually active woman to use adequate contraceptive methods.
4. Active medical illness which might make participation hazardous, such as untreated hypertension, hepatitis with SGOT or SGPT > 3 times normal, unstable diabetes.
5. Active psychiatric disorder which might interfere with participation or make participation hazardous, including DSM-IV schizophrenia, bipolar disorder with mania or psychosis, and depressive disorder with suicide risk or 1 or more suicide attempts within the past year.
6. Physiologically dependent on alcohol or sedative-hypnotics with impending withdrawal. Other substance use diagnoses are not exclusionary. Multiple substance use is common in this population, and such an exclusion would rule out a large proportion of the population and limit the generalizability of the study.
7. History of allergic reaction to buprenorphine, naltrexone, naloxone, clonidine, or clonazepam.
8. Chronic organic mental disorder (e.g. AIDS dementia).
9. History of accidental drug overdose in the last 3 years as defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.
10. Currently receiving any other investigational drug, or has used any other investigational drug within 30 days of study entry.
11. Currently prescribed or regularly taking opiates for chronic pain or medical illness or those individuals anticipating surgical procedures which will necessitate opioid medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Nunes, M.D., Study Director — Columbia University; Maria Sullivan, M.D., Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- See also: Information on the Substance Treatment and Research Service — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Depot Naltrexone: Depot Naltrexone. Vivitrol (380 mg)given monthly depot naltrexone: On the afternoon of Day 7, patients assigned to Depot-BNT receive an intramuscular injection of Vivitrol (380 mg) in one buttock. The patient spends the night of Day 7 in the hospital and is discharged on the morning of Day 8. Each injection contains 192 mg of naltrexone. The double dose (384 mg) is what was found to produce optimal blockade and outcome in preliminary work. During the subsequent 6-month course of outpatient treatment, patients are dosed with two injections (384 mg total) of depot naltrexone at monthly intervals (weeks 4, 8, 12, 16, 20).
Period: Overall Study
Arm/Group | Depot Naltrexone | Oral Naltrexone
Started | 28 | 32
Completed | 16 | 9
Not Completed | 12 | 23
Not completed — Stopped attending study visits | 9 | 11
Not completed — Continued opioid use | 3 | 2
Not completed — Non-compliance with study meds | 0 | 3
Not completed — Refused Oral Naltrexone | 0 | 1
Not completed — Moved out of state | 0 | 1
Not completed — Scheduling Issues | 0 | 3
Not completed — Death | 0 | 1
Not completed — Psychiatric hospitalization | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Depot Naltrexone | Oral Naltrexone | Total
Number analyzed (Participants) | 28 | 32 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 32 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 24 | 26 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 21 | 38
  Hispanic | 4 | 9 | 13
  Black | 5 | 2 | 7
  Asian | 1 | 0 | 1
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 32 | 60

OUTCOME MEASURES:

1. Primary Outcome: Treatment Retention
Description: compliance with being retained in treatment protocol
Time Frame: over the course of 24 weeks or length of study participation
Measure: Count of Participants; unit: Participants
Arm/Group | Depot Naltrexone | Oral Naltrexone
Number analyzed (Participants) | 28 | 32
Participants
  4 Weeks | 24 | 20
  12 Weeks | 17 | 14
  24 Weeks | 16 | 9

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Depot Naltrexone | Oral Naltrexone
Serious Adverse Events (participants affected / at risk) | 6/28 | 3/32
Other Adverse Events (participants affected / at risk) | 16/28 | 25/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Depot Naltrexone (N=28) | Oral Naltrexone (N=32)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
chest pain (Vascular disorders) | 0 (0) | 1 (1)
Spontaneous abortion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
increased anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Cannabis induced psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Cardiac death (Vascular disorders) | 0 (0) | 1 (1)
car accident (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Depot Naltrexone (N=28) | Oral Naltrexone (N=32)
Insomnia (Psychiatric disorders) | 7 (7) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 6 (6)
Anxiety (Psychiatric disorders) | 5 (5) | 5 (5)
depression (Psychiatric disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No